CLINICAL TRIAL: NCT01432249
Title: Post Marketing Surveillance To Observe Safety And Efficacy Of Enbrel In Pediatric Patients With Psoriasis
Status: Withdrawn | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801135
Record Dates: First submitted 2011-08-05; First posted 2011-09-12 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Pediatric Psoriasis
Keywords: pediatric psoriasis; enbrel; safety; efficacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Enbrel: The patients who are prescribed Enbrel for pediatric psoriasis
  Interventions: Drug: Enbrel group

INTERVENTIONS:
Drug: Enbrel group — will be decided by treating physicians

SUMMARY:
Enbrel was first approved as new medicine on 06 Oct 2003 in Korea and the indication of Pediatric Psoriasis was approved on 23 Sep 2009. However, as required for any new indication approved by Korea Food and Drug Administration (KFDA), safety and efficacy information of new indication should be provided at minimum 600 subjects administered in the setting of routine practice during the initial 4 years after new indication approved.

DETAILED DESCRIPTION:
All patients enrolled should meet the usual prescribing criteria for Enbrel in psoriasis as per the local product information for usage.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents aged 8 years to 17 years at time of consent
2. Chronic severe psoriasis patients who are inadequately controlled by, or are intolerant to, other systemic therapies or phototherapies

Exclusion Criteria:

1. Patients with known hypersensitivity to Enbrel or any component of the product
2. Patients with active infections including chronic or localized infections such as tuberculosis (Treatment of Enbrel should not be initiated)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients (ages of 8~17)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Safety measured by discontinuation due to adverse events | 6 month

SECONDARY OUTCOMES:
Proportion of subjects achieving a status on the PGA (Physician's Global Assessment) of psoriasis of clear (0), clear/almost clear (0/1), or clear/almost clear/mild (0/1/2) at 12 weeks and 24 weeks | 6 month
Proportion of subjects achieving a 50% and 75% improvement from baseline in PASI (Psoriasis Area-and-Severity Index) over 12 weeks and 24 weeks | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801135&StudyName=Post%20Marketing%20Surveillance%20To%20Observe%20Safety%20And%20Efficacy%20Of%20Enbrel%20In%20Pediatric%20Patients%20With%20Psoriasis